CLINICAL TRIAL: NCT00183859
Title: Phase I Clinical and Pharmacokinetic Trial of Intra-Peritoneal Irinotecan
Brief Title: Clinical and Pharmacokinetic Trial of Intra-Abdominal Irinotecan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0C-99-7
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Adenocarcinoma; Gastric Cancer
Keywords: solid tumor; phase I; phase one
MeSH Terms: conditions — Adenocarcinoma; Stomach Neoplasms | interventions — Irinotecan

ARMS (1):
- A (Experimental): Intraperitoneal Irinotecan
  Interventions: Drug: irinotecan

INTERVENTIONS:
Drug: irinotecan — Intraperitoneal Irinotecan given every three weeks

SUMMARY:
This is a research study for patients that have an advanced cancer that is confined mostly to the abdominal cavity and have failed treatment with conventional therapy, or for which no standard treatment exists. The purpose of this study is to determine the dose of a chemotherapy drug (called irinotecan) that can be administered safely into the abdominal cavity. We also wish to identify the side effects of irinotecan when it is administered directly into the abdomen. In this study, we will also determine the levels of irinotecan in the blood and in the abdominal cavity.

Irinotecan is a chemotherapy drug that can decrease the size of several different tumors. It is approved by the FDA for the treatment of colon cancer. It appears that some other chemotherapy drugs are more effective and may have less side effects when they are administered directly into the abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent, metastatic, or residual cancer with disease confined mostly to the peritoneal cavity. Patients with asymptomatic extra-peritoneal disease are eligible.
* Measurable or evaluable disease. Patients with malignant ascites or carcinomatosis only (documented by cytology or during surgery) are eligible. Patients with ovarian cancer and disease manifested only by an elevated CA-125 are also eligible.
* Adequate hepatic, renal, and bone marrow functions: bilirubin less than or equal to 2.0 mg/dl; creatinine less than or equal to 2.0 mg/dl, alkaline phosphatase less than or equal to 3 x upper limit of normal (uln), AST or ALT less than or equal to 3 x uln; AGC greater than or equal to 1500, platelets greater than or equal to 100,000.
* SWOG performance status 0-2
* Fully recovered from acute toxicities from prior surgery, chemotherapy, or radiation therapy.
* Patients must use an approved method of birth control.

Exclusion Criteria:

* Medical, social, or psychological factors which could prevent patient from receiving treatment.
* Prior therapy with intra-peritoneal irinotecan
* Significant intra-peritoneal adhesions detected clinically or by prior surgical exploration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 1999-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose (MTD) of irinotecan when administered by an intra-peritoneal route every three weeks. | 6 weeks

SECONDARY OUTCOMES:
To determine the pharmacokinetics of intra-peritoneal irinotecan. | One day
To determine the toxicity profile of intra-peritoneal irinotecan. | 30 days after patient receives last dose

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, M.D., Principal Investigator — U.S.C. / Norris Comprehensive Cancer Center
Locations (1):
- U.S.C. / Norris Comprehensive Cancer Center, Los Angeles, California, United States